CLINICAL TRIAL: NCT01706562
Title: Retrospective Observation of Empirical Antifungal Therapy With Itraconazole
Brief Title: A Study of Empirical Antifungal Therapy With Itraconazole
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR017839; ITRFUN4055 (Other: Janssen Korea, Ltd., Korea); ITR-KOR-5088 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Neutropenia
Keywords: Neutropenia; Hematologic malignancy; Itraconazole; Fungal infection; Antifungal agent; Neutropenic fever
MeSH Terms: conditions — Neutropenia; Hematologic Neoplasms; Mycoses; Febrile Neutropenia | interventions — Itraconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Itraconazole
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — Itraconazole intravenous (IV) 200 mg twice daily for 2 days, a total of 4 doses and then 200 mg once daily until clinically significant resolution of neutropenia.

SUMMARY:
The purpose of this study is to investigate the overall success rate of itraconazole intravenous treatment for a period of more than 7 days.

DETAILED DESCRIPTION:
This is a retrospective study ie, a study that looks backward in time, usually using medical records and interviews with patients who are already known to have a disease, in patients with itraconazole intravenous prescription as an empirical (based on practical experience) antifungal agent. This study collects baseline information about underlying disease, sign of fungal infection, neutropenia (a decrease in white blood cells), neutropenic fever duration and the reason for discontinuation. Neutropenia is defined as a neutrophil (white blood cell) count of ≤500 cells/mm3 or a count of ≤1000 cells/mm3 with a predicted decrease to ≤500 cells/mm3. Fever is defined as a body temperature ≥38.3 Celsius degrees at least once a day with no definite external factor or a body temperature of ≥38 Celsius degrees continued for at least 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neutropenic fever who receive therapy for inhibiting or preventing development of neoplasms (abnormal growth of tissue) or stem cell transplantation (stem cell is a cell whose daughter cells may differentiate into other cell types) for hematologic malignancies (cancers that affect blood, bone marrow and lymph nodes)
* Patients who receive itraconazole intravenous (IV) treatment for more than 7 days

Exclusion Criteria:

* Childbearing women who are pregnant or likely to be pregnant during the study period and men who are neither infertile nor willing to refrain from sexual relations but whose partner does not conduct an effective contraception
* Fever due to documented fungal infection
* Hepatic dysfunction
* Kidney abnormalities
* Patients who are not eligible for the study participation based on warnings, precautions and contra medications in the package insert of the study drug at the investigator's discretion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of patients with hematologic malignancy who visited a study center and were treated with itraconazole intravenous (IV) for more than 7 days.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Success rate of itraconazole treatment when used for more than 7 days | From 7 days to approximately 2 weeks
  Treatment success is achieved when neutropenia is resolved, ie, when the blood cells count is within the normal reference range.

SECONDARY OUTCOMES:
Success rate of itraconazole treatment until neutropenia is resolved | Approximately 2 weeks
  Treatment success is achieved when neutropenia is resolved, ie, when the blood cells count is within the normal reference range.
Drop out rate due to the lack of efficacy of itraconazole treatment | Approximately 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea